CLINICAL TRIAL: NCT00107666
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Proof of Concept Clinical Study of CTI-01 in Patients Undergoing Major Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: CTI-01 (Ethyl Pyruvate) Safety and Complication Prevention in Cardiac Surgery Patients on Cardiopulmonary Bypass (CPB)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Critical Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTI-01-C04-201
Record Dates: First submitted 2005-04-06; First posted 2005-04-07 (Estimated); Last update posted 2006-03-17 (Estimated); Status verified 2006-03

CONDITIONS: Coronary Disease; Heart Valve Diseases
Keywords: Coronary artery bypass grafting; Heart valve prosthesis implantation; Cardiopulmonary bypass; Oxidative stress; Inflammation; Endotoxemia
MeSH Terms: conditions — Coronary Disease; Heart Valve Diseases; Inflammation; Endotoxemia | interventions — ethyl pyruvate

INTERVENTIONS:
Drug: CTI-01 (ethyl pyruvate)

SUMMARY:
Over 500,000 patients undergo cardiac surgery with CPB in the United States annually. Although mortality rates have decreased with advances in perioperative care, many patients are affected by postoperative organ dysfunction. The incidence of complications may exceed 30%. It has been speculated that an exaggerated inflammatory response to surgical trauma and the CPB machine are likely causes for this morbidity. Factors predisposing organ dysfunction include tissue injury, endotoxemia, and oxidative stress. High risk patients can be identified preoperatively through the validated Parsonnet Additive Risk Score. CTI-01 has demonstrated potent anti-inflammatory and tissue protection activity in multiple animal models of disease including pancreatitis, ischemia-reperfusion injury, sepsis, renal injury, and endotoxemia. These findings support its clinical use in critical care medicine including cardiac surgery. Patients will receive a total of six doses, administered intravenously just prior to and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Parsonnet additive risk score greater than or equal to 15
* Scheduled CABG (coronary artery bypass grafting) and/or cardiac valve repair or replacement surgery using cardiopulmonary bypass

Exclusion Criteria:

* Emergency cardiac surgery
* Significant concomitant surgery
* Minimally invasive or thoracic surgical approach
* Preoperative mechanical assist device
* Body weight <50 kg or >140 kg
* Active systemic infection
* Creatinine >3.0 mg/dL
* History of hematologic or coagulation disorders
* History of malignancy (past year)or organ transplantation
* Use of immunosuppressive drugs or current immunosuppressed condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-04; Study Completion 2006-04

PRIMARY OUTCOMES:
Death
Composite morbidity endpoint

SECONDARY OUTCOMES:
Respiratory dysfunction
Cardiac dysfunction
Renal dysfunction
Gastrointestinal dysfunction
Mental status
Length of ICU (Intensive Care Unit)/hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Walter Newman, Ph.D., Study Director — Critical Therapeutics Incorporated
Locations (17):
- United States (17):
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - University of Southern California, Los Angeles, California
  - Kaiser Permanente, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Research Support Personnel, Wichita, Kansas
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - NYU Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University - Brody School of Medicine, Greenville, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Chester County Hospital - The Cardiovasular Center, West Chester, Pennsylvania
  - St. Luke's Episcopal Hospital/Texas Heart Institute, Houston, Texas
  - MultiCare Health System, Tacoma, Washington
  - Medical College of Wisconsin - VA Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Background] Parsonnet V, Dean D, Bernstein AD. A method of uniform stratification of risk for evaluating the results of surgery in acquired adult heart disease. Circulation. 1989 Jun;79(6 Pt 2):I3-12. PMID 2720942
- [Background] Bennett-Guerrero E, Ayuso L, Hamilton-Davies C, White WD, Barclay GR, Smith PK, King SA, Muhlbaier LH, Newman MF, Mythen MG. Relationship of preoperative antiendotoxin core antibodies and adverse outcomes following cardiac surgery. JAMA. 1997 Feb 26;277(8):646-50. PMID 9039883
- [Background] Ulloa L, Ochani M, Yang H, Tanovic M, Halperin D, Yang R, Czura CJ, Fink MP, Tracey KJ. Ethyl pyruvate prevents lethality in mice with established lethal sepsis and systemic inflammation. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12351-6. doi: 10.1073/pnas.192222999. Epub 2002 Sep 3. PMID 12209006
- [Background] Woo YJ, Taylor MD, Cohen JE, Jayasankar V, Bish LT, Burdick J, Pirolli TJ, Berry MF, Hsu V, Grand T. Ethyl pyruvate preserves cardiac function and attenuates oxidative injury after prolonged myocardial ischemia. J Thorac Cardiovasc Surg. 2004 May;127(5):1262-9. doi: 10.1016/j.jtcvs.2003.11.032. PMID 15115981
- [Background] Fink MP. Ethyl pyruvate: a novel anti-inflammatory agent. Crit Care Med. 2003 Jan;31(1 Suppl):S51-6. doi: 10.1097/00003246-200301001-00008. PMID 12544977